CLINICAL TRIAL: NCT04964245
Title: Respiratory Measurement of Volume Change Using Accelerometer, Thermographic Camera Electrical Impedance Tomography and Motion Correlation Analysis Using Mattress Sensor in Healthy Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4-2020-1320
Record Dates: First submitted 2021-07-01; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Healthy Adult
Keywords: Respiration; Tidal volume
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiration monitoring group (Experimental): The respiration is simultaneously measured by accelerometer, thermographic camera, Impedance Tomography, and mattress sensor.
  Interventions: Device: accelometer; Device: thermographic camera; Device: Electrical Impedance Tomography; Device: Mattress Sensor

INTERVENTIONS:
Device: accelometer — the respiration parameters are measured using an accelometer.
Device: thermographic camera — the respiration parameters are measured using an thermographic camera.
  Other Names: FLIR 655sc
Device: Electrical Impedance Tomography — the respiration parameters are measured using an electrical impedance tomograhy.
Device: Mattress Sensor — the respiration parameters are measured using an Mattress pressure

SUMMARY:
Tidal volume can be the most important technical indicator for ventilation. Measuring the volume of breathing can be used as an indicator of how effective a patient's gas exchange is, and as a predictive indicator of the statue of respiratory disease indirectly. These Tidal volumes can be measured using spirometry and pneumotachograph, and the breathing volume and the rate of airflow can directly or indirectly evaluate the lung function of the patient.

However, spirometry has limitations that patients who are difficult to measure, and that it is difficult to measure in bed. In this work, the movement of the thorax due to breathing is measured in a non-invasive manner (accelerometer, thermographic camera) and the accuracy is compared through changes in thoracic impedance obtained through Pulmovista 500. Furthermore, we would like to correlate the motion of the measured object through a mattress sensor.

ELIGIBILITY:
Inclusion Criteria:

1. over 19, under 50 years old and common BMI
2. non-smoking, person without cardiopulmonary disease.

Exclusion Criteria:

1. smoking, cardiopulmonary, infectious diseases.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
The accuracy of respiration measurements | about 20 min
  The accuracy respiration measurements between thermographic camera, accelerometer, electrical impedance tomography, and mattress sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Jeongmin Kim, Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided